CLINICAL TRIAL: NCT02427919
Title: The DEtection of G-CSF REceptor With Flow Cytometry and Identification of the Effect of G-CSF After Salvage Chemotherapy in Relapsed or Refractory AML
Brief Title: Granulocyte Colony Stimulating Factor (G-CSF) After Salvage Chemotherapy in Refractory AML
Acronym: DeGREE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Jae-Ho, Yoon, Clinical assistant professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHSCTC-R02-DeGREE
Record Dates: First submitted 2015-04-17; First posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: G-CSF; G-CSF receptor; AML; refractory AML; Neutropenic fever; salvage chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Febrile Neutropenia | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early G-CSF use (Experimental): Refractory AML undergoing salvage chemotherapy (MEC regimen in AML). After finishing application of chemotherapy, G-CSF will be started post chemotherapy D+7~D+10 when blasts disappear from peripheral blood smear.
  When blasts reappear on peripheral blood smear, G-CSF will be discontinued.
  Intervention type : Drug Intervention name : G-CSF (Filgrastim)
  -> Comparison of the effect of G-CSF (Filgrastim) use
  Interventions: Drug: G-CSF
- No or delayed G-CSF use (Active Comparator): Refractory AML undergoing salvage chemotherapy (MEC regimen in AML). After finishing application of chemotherapy, G-CSF will not be applied at least post chemotherapy D+25~D+28. If patient suffers from severe infectious complication and when no blasts are detected on peripheral blood smear, G-CSF can be started then.
  Intervention type : Drug Intervention name : G-CSF (Filgrastim)
  -> Comparison of the effect of G-CSF (Filgrastim) use
  Interventions: Drug: G-CSF

INTERVENTIONS:
Drug: G-CSF — Comparison of the effect of G-CSF use
  Other Names: Filgrastim

SUMMARY:
Granulocyte Colony Stimulating Factor (G-CSF, filgrastim) is now widely used after chemotherapy which complicates hematological toxicity involving neutropenia. As prolonged neutropenia leads to neutropenic fever due to bacteremia or fungal infection, the use of G-CSF prevents severe infectious complication in various cancer patients.

In acute myeloid leukemia (AML), leukemic blasts have been expected to have G-CSF receptor which may be stimulated by G-CSF, and refractory patients were not treated with G-CSF in salvage chemotherapy in Catholic blood and marrow transplantation (BMT) Center for a long time. This strategy induced prolonged neutropenia and a lot of infectious complications some of which led to deaths.

Although there are some data which remind us G-CSF may proliferate leukemic blasts, the investigators also identified several reports which suggested that subgroup with G-CSF use showed acceptable CR rate and improved survival outcomes compared to a subgroup without G-CSF use.

Therefore investigators are now trying to identify the effects of G-CSF for refractory AML patients in salvage chemotherapy setting regarding the duration of neutropenia and admission, incidence of infectious complications and the duration of antibiotics application. Furthermore, overall response rate (CR+CRi) after salvage chemotherapy and survival outcomes will be calculated according to G-CSF use.

Also, investigators will detect G-CSF receptor using cluster of differentiation 114 (CD114), and analyze the clinical outcomes according to the subgroups with or without using G-CSF during neutropenic period.

DETAILED DESCRIPTION:
Patients will be treated with mitoxantrone and etoposide and cytarabine. Patients will be randomly divided according to the usage of G-CSF.

Subgroup with G-CSF will be treated with G-CSF after 7~10 days post-chemotherapy, when blasts will disappear from peripheral blood.

Subgroup without G-CSF will be observed until 25~28 days post-chemotherapy. If blood counts are nor recovered, the investigators can perform bone marrow biopsy to identify the status of the bone marrow.

After then, G-CSF can be applied if blasts are not observed in both peripheral blood and bone marrow.

When absolute neutrophil counts are recovered and there are no evidence of infectious complications, patients will discharge safely from hospital.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0~2
* AML with remission failure after standard chemotherapy
* Stable liver and renal function (=< Upper normal limit (UNL) x 2.5)
* Stable heart and lung function (Ejection Fraction (EF) > 45%, Forced expiratory volume at one second (FEV1) > 40%)

Exclusion Criteria:

* Acute promyelocytic leukemia
* Central nervous system (CNS) involvement
* Uncontrolled bleeding
* Uncontrolled infectious complication
* Pregnancy, Breast feeding
* Significant cardiovascular disease within 6 months
* Significant organ failure (> UNL x 2.5)

Ages: 17 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Recovery time from neutropenia | 30 days

SECONDARY OUTCOMES:
Incidence of neutropenic fever and infectious complication | 30 days
Complete remission rate | 45 days
Overall survival | 3 year
Disease free survival | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Ho Yoon, Study Chair — Catholic BMT Center, Seoul St Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, Banpodaero 222, South Korea